CLINICAL TRIAL: NCT07311759
Title: Safety and Efficacy of Intralesional 0.5% Triamcinolone Acetonide in 0.2% Fluconazole Solution vs 0.1% Topical Mometasone Furoate With 2% Miconazole Nitrate Cream in the Treatment of Chronic Paronychia: An Intraindividual Randomized Controlled Trial.
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basant Ahmed Mohamed Abdelaal Helal, Dermatology Specialist, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-255-2024
Record Dates: First submitted 2025-08-05; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-11

CONDITIONS: Chronic Paronychia
Keywords: Intralesional triamcinolone; Chronic paronychia; Intralesional fluconazole
MeSH Terms: interventions — Fluconazole; Mometasone Furoate; Miconazole

STUDY DESIGN:
Intervention Model Description: The affected fingernails in each patient are randomized, by simple randomization technique, to either receive intralesional or topical treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralesional Triamcinolone acetonide and fluconazole (Active Comparator): The proximal nail fold is cleansed with alcohol. Triamcinolone acetonide and fluconazole in the ratio of 1:7, yielding a triamcinolone acetonide concentration of 5mg/ml, is injected through the affected nail fold with a 30-gauge, 1-mL insulin syringe needle. The nail fold is divided into 2 halves and a maximum of 0.5 cc is injected in both halves or till there is swelling /edema of the nailfold. Injections are administered every 4 weeks until the end of treatment response, or for a maximum of 3 months
  Interventions: Drug: Intralesional triamcinolone acetonide and fluconazole
- Topical treatment with mometasone furoate and miconazole nitrate (Active Comparator): Topical treatment in the form of twice daily application of combined steroid and antifungal (mometasone furoate and miconazole nitrate, Elica-M®) till the end of treatment response or for a maximum of 3 months.
  Interventions: Drug: Topical mometasone furoate and miconazole nitrate, Elica-M®

INTERVENTIONS:
Drug: Intralesional triamcinolone acetonide and fluconazole — Triamcinolone acetonide and fluconazole in the ratio of 1:7, yielding a triamcinolone acetonide concentration of 5mg/ml, is injected through the affected nail fold with a 30-gauge, 1-mL insulin syringe needle.
  Arms: Intralesional Triamcinolone acetonide and fluconazole
Drug: Topical mometasone furoate and miconazole nitrate, Elica-M® — Topical treatment in the form of twice daily application of combined steroid and antifungal (mometasone furoate and miconazole nitrate, Elica-M®) till the end of treatment response or for a maximum of 3 months.
  Arms: Topical treatment with mometasone furoate and miconazole nitrate

SUMMARY:
Our objective is to compare the efficacy and safety of intralesional corticosteroids + fluconazole solution to corticosteroid with an antifungal topical preparation, in the management of chronic paronychia.

DETAILED DESCRIPTION:
Chronic paronychia (CP) is defined as inflammation of the nail fold(s) of more than 6 weeks duration (Shafritz and Coppage, 2014). It is now considered as a form of hand eczema, caused primarily by irritation of the nail folds by environmental allergens. This leads to recurrent inflammation of nail folds, followed by fibrosis and inability to generate the cuticle, ending in loss of the waterproof seal, moisture retention, and compromise of blood supply due to fibrosis. These can explain why CP is commonly resistant to topical and even systemic treatments. Candida infection is thought to be a secondary event in a subset of cases (Relhan and Bansal, 2022), with positive fungal culture in about 56.1% of cases (Bahunuthula et al., 2015) Important risk factors for the development of CP include occupations with excessive exposure to moisture and irritants (e.g. housewives, cooks, and health care providers), immunosuppression (e.g. diabetes mellitus and HIV); due to increased risk of secondary colonization, and some medications (e.g. retinoids) (Relhan and Bansal, 2022). A higher incidence of contact sensitization and Candida hypersensitivity in these patients has been reported, (Bahunuthula et al., 2015) thus candidal control may be of help to ameliorate the disease.

Clinically, CP presents with erythema, pain and swelling of one or more of the nail folds for >6 weeks. It generally affects multiple fingernails, more commonly, of the dominant hand. Nail matrix may be secondarily affected leading to transverse ridging, discoloration, Beau's lines, or onychomadesis (Shafritz and Coppage, 2014, Atiş et al.,2018). The last updated severity scale for CP has been proposed in 2018, taking into account the number of affected nail folds, erythema, edema, nail plate and cuticle changes (Atiş et al.,2018).

Management of CP relies mainly on avoidance of the irritants and topical corticosteroids which are now considered the mainstay of treatment (Shafritz and Coppage, 2014). Systemic antifungals are used in cases with associated candida infection (Tosti et al., 2002).

Intralesional steroid injection, in the form of monthly injections of triamcinolone acetonide (2.5- 10 mg/mL), is used for the treatment of nail psoriasis, nail lichen planus and twenty-nail dystrophy. It is, however, scarcely mentioned in literature in the management of CP (Baran, 2001). In addition, the optimal treatment regimen and injection technique have not yet been established, and no recent relevant studies exist.

Surgical treatment is reserved for cases of CP of more than 6-month duration, that has been resistant to medical treatment (Relhan et al., 2014)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic paronychia affecting ≥ 2 fingernails in the dominant hand.
2. Patients not receiving any relevant systemic treatment for at least 4 weeks before initiation of our study
3. Patients not receiving any relevant topical treatment for at least 2 weeks before initiation of our study

Exclusion Criteria:

1. Patient with peripheral vascular disease or Raynaud's phenomenon
2. Pregnant and lactating females
3. Patients with autoimmune diseases e.g., connective tissue diseases, psoriasis, reactive arthritis, and pemphigus.
4. Patients with solid or hematological malignancies.
5. Patients on systemic drugs that are known to cause chronic paronychia e.g. retinoids.
6. Patients with any visible focus of infection at the injection site or in the vicinity, including patients with superimposed attack of acute paronychia.
7. Onychomycosis or any associated nail disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Comparison between the chronic paronychia severity index scale before and after treatment in each group | 4 months
  Evaluation of proximal and lateral nail fold involvement, edema, erythema, nail plate changes and cuticle involvement for each affected nail before and after treatment using the chronic paronychia severity index score according to Atis et al, 2018 to measure the efficacy of each group on its own
Comparison of the change in chronic paronychia severity index scale between both groups | 4 months
  According also to Atis et al, 2018. We will grade the affected nails using the chronic paronychia severity index scale and measure the difference between before and after treatment between both groups, where pre-treatment evaluation to check for any bias and post-treatment to check which intervention was more superior.
Comparison of percentage of patients who achieved complete response (chronic paronychia severity index scale =0) between both groups. | 4 months
  We will assess whether the patient had a complete response or not according to the chronic paronychia severity index scale equals to zero

CONTACTS AND LOCATIONS:
Overall Officials: Yousra A Azzazi, Lecturer of Dermatology, Study Director — Cairo University; Mohamed M El-Komy, Professor of Dermatology, Study Chair — Cairo University; Habiba K Edrees, Dermatology Resident, Principal Investigator — Cairo University; Khadija A Affify, Dermatology resident, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT07311759/Prot_SAP_000.pdf